CLINICAL TRIAL: NCT04148469
Title: Benefits and Harms of Dry Needling vs Transcutaneous Nerve Stimulation and Dry Needling in Patients With Chronic Myofascial Neck Pain and Relationship With Psychological Influences
Brief Title: Dry Needling Effectiveness and Post-punction Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: urjc20-13
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Neck Pain
Keywords: Miofascial pain syndrom.; Trigger point.; Dry needling.; Transcotaneous Nerve Stimuilation.; Hipoalgesia
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- dry needling and TENS (Experimental): A dry needling treatment was performed on trapezius trigger point number 2, and just after thar, a TENS curretn was applied. Patients will be reassed on fourth day after treatment.
  Interventions: Procedure: Transcutaneous Nerve Stimulation.
- Placebo (Placebo Comparator): A placebo dry needling was performed on trapezius trigger point number 2. Patients will be reassed on fourth day after treatment.
  Interventions: Procedure: Placebo needling
- dry needling (Experimental): A dry needling treatment was performed on trapezius trigger point number 2. Patients will be reassed on fourth day after treatment.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Dry needlin is a manual therapy technique used for miofascuial pain syndrom treatment. The patient will be supine, in a confortable position. The therapist localizes the trapezius trigger point number 2 and then performes the needling until 2 REL are obtenined. The patient will remain supine during 15 minutes.
  Arms: dry needling
Procedure: Transcutaneous Nerve Stimulation. — Transcutaneous Nerve Stimulation (TENS) is a current used for pain treatment. The needle will be used as the negative pole and a adhesive patch 2 centimeters lateral will be the positive pole. The frecuency selected will have 2 Hz with pulses of 120 microseconds. The currente will be applied for 15 minutes.
  Arms: dry needling and TENS
Procedure: Placebo needling — No active technique is performed with the placebo needling. Patient will be supine and a placebo needle willb be performed. The patient will remain supine for 15 minutes.
  Arms: Placebo

SUMMARY:
The purpose of this estudy was to dertermine if the application of Transcutaneous Nerve Stimiulation (TENS) current have an hypoalgesic effect on pattientes suffering from miofascial neck pain, compared with a only dry needling treatment. Psicological varaibles were also mesured in order to determine how they change after each treatment.

DETAILED DESCRIPTION:
All patients suffered from mechanical neck pain and were randomized into three groups of treatment. A doible blinded control was carryed out. The main outcome messures were Visual Analogue Scale (VAS). The scondary outcome messures were Pressure Pain hreshold (PPT) and Active Range of Movement (ROM). Also psicologicla messures were taken, like Neck Dissability Index, Level of stress and ansiety, Fear Pain and Pain Avoidance Strategies.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical Neck pain of at least 6 months.
* VAS 2 or greather.
* Existance of miofascial trigger point in trapezius muscle assesed by an expert PT.

Exclusion Criteria:

* Neck pain due secondary to ostheoporosis, metastasis, neoplasias, fractures, infections, cervical stenosis or infexious procces.
* Headache secondary to medular compression presenting one o the following signs: abnormal sensitivity, hiperreflexia, clonus, spread weakness, cervical hernia.
* Neck pain with radiculopathy.
* Whiplash.
* Vertebrobasilar syndrome.
* Dizzyness.
* Pregnancy.
* Having received dry needling treatment before.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-06-12 (Actual); Study Completion 2013-12-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Patients will be reassed in four days.
  Visual Analogue Scale (VAS) is a subjective evaluation. There are previous studies that demonstrate its reliability and its sensitivity, wich give validity to VAS messures. The messure is made using a two sides 10 centimeters scale. The patient´s face shows an increasing slope that allows the patient to mark his pain level. That mark has his equivalent number on the scale, so 0 is no pain and 10 is maximum pain. A differece of 2 points on the scale means the minimum clinically significant change.

SECONDARY OUTCOMES:
Active Cervical Range of Movement | Patient will be reassed in four days.
  To messure the cervical range of movement, a CROM will be used. The CROM is a special goniometer that allows therapists to messure cervical movements. It conists on trhee pairs of inclinometers that allow reserchers to messure range of flexion-extension, lateral flexion and rotation. The CROM has a porved reliability, providing a inter-meter reliability from 0,7 to 0,9 and an intra-meter reliability from 0,8 to 0,87. The patient will be seated on a cheir, and he´ll perform cervical movements actively, just untill he starts to feel his pain. Each movement will be messure three times, and the average will be taken.
Pressure Pain Threshold | Patients will be reassed in four days.
  Pressure Pain Threshold (PPT) is the minimun pressure needed to araise pain. To messure PPT, an digital algometer will be used. An algometer consists on a 1 square centimeter rubber piece inserted on a pressure gauge. Previous studies have shown the reliability of this method (ICC=0,91) and also inter meter (ICC from 0,82 to 0,97) and intra meter (ICC=0,78). The minimun detectable change on the cervical area goes from 0,44 Kg/cm2 to 1,11 Kg/cm2. We will apply the algometer over trapezius trigger point number 2, and the patient will tell the therapist when he start to feel hgis pain. We´ll do the messure 3 times and the average will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Vicente León Hernández, PT, Principal Investigator — Universitdad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain